CLINICAL TRIAL: NCT06943560
Title: Emotion Regulation Selection Flexibility Training for PTSD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Gal Sheppes, Principal Investigator of Emotion Regulation Lab, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sheppes01
Record Dates: First submitted 2025-03-02; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: PTSD
Keywords: EMOTION REGULATION
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Emotional Regulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regulatory selection Flexibility Training (Experimental)
  Interventions: Behavioral: Emotion Regulation Selection Flexibility Training
- Tight Active control Training (Experimental)
  Interventions: Behavioral: Emotion Regulation Active control Training

INTERVENTIONS:
Behavioral: Emotion Regulation Selection Flexibility Training — 7 online computerized regulatory selection training sessions that includes a fully computerized part, and an interactive, human operated part guided by a clinician and home assignments between intervention session to be completed on days without sessions. Psychoeducation includes information on selection of appropriate strategy according to the regulatory selection flexibility rule (i.e., distraction for high intensity vs reappraisal in low intensity). In the computerized task participants are exposed to emotional words and are asked to select a regulatory strategy in a flexible matter according to the regulatory selection flexibility rule, and receive feedback on whether they chose flexibly or not. Following , they are instructed to implement the chosen strategy. Homework includes choosing two daily events one of high intensity and a second one of low intensity, and describe which strategy they selected and how they implemented their chosen strategy according to the flexibility rule.
  Arms: Regulatory selection Flexibility Training
Behavioral: Emotion Regulation Active control Training — All the interventional sections are similar to the experimental group except that in the control group we omit the regulatory selection rule that defines which strategy is compatible with which emotional situation.
  7 online computerized regulatory selection training sessions that includes a fully computerized part, and an interactive, human operated part guided by a clinician and home assignments between intervention session to be completed on the days without sessions. Psychoeducation explicitly included information on regulatory strategies (without the regulatory selection flexibility rule). In the computerized task participants are exposed to the same emotional words and are asked to choose freely a regulatory strategy (without the regulatory selection flexibility rule or feedback), and implement it. Homework includes choosing two daily events and selecting and implementing a regulatory strategy (without the regulatory selection flexibility rule).
  Arms: Tight Active control Training

SUMMARY:
This clinical study will examine the efficacy of a novel intervention aimed at improving Regulatory Selection Flexibility and PTSD symptoms among adult individuals with PTSD symptoms, compared to a tight active control group.

DETAILED DESCRIPTION:
Regulatory Selection Flexibility is defined as the ability to select regulatory strategies according to differing situational demands (i.e., regulatory selection flexibility rule; distraction for high intensity vs reappraisal in low intensity). The main questions it aims to answer are: [1] Can PTSD individuals improve Regulatory Selection Flexibility [2] Does improved Regulatory Selection Flexibility associate to reduction in PTSD symptoms? Participants will be randomly assigned to either a Flexibility Training or a closely matched Active regulatory selection Control Training group. Participants in both groups will receive a novel online bi weekly seven session intervention which is matched on all aspects of the intervention except for the flexibility rule as follows, the intervention consists of three modules: (a) Psychoeducation; both groups receive information on regulatory strategies (distraction and reappraisal). The test group includes explicit psychoeducation on appropriate strategy selection according to the regulatory selection flexibility rule. (b) Computerized Regulatory Selection Task; both groups are exposed to high and low negative intensity emotional words and are asked to select a regulatory strategy. Only the test group receives the flexibility rule and its application via feedback. (c) Two homework task for between sessions. Both groups are instructed to choose two daily events and report which regulatory strategy they chose and implemented. The test group is instructed to choose a high and low intensity event and implement flexible selection. Each session begins with a brief overview on their home task, followed by corrective feedback in test group when necessary.

Primary outcome measures were acquired via the computerized assessment of Regulatory Selection Flexibility Paradigm and clinical questioners for PTSD symptoms pre, immediately post and at 3-month post intervention follow up.

To examine the efficacy of the regulatory selection intervention and its clinical effects, according to a-priori power analysis and expected drop out of 20%, 80 participants that meet me PTSD cutoff will be enrolled and randomly assigned to one of two conditions: Experimental group (Regulatory Selection Flexibility Training) or active control (Regulatory Selection without Flexibility Training).

Following intervention, the investigators expect that (a) Both groups will show PTSD symptom reduction. (b) That relative to the active control group, the experimental group will show improvement in regulatory selection flexibility pre-to-post intervention, and (c) That relative to the active control group, the experimental group will show greater reduction in PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* native Hebrew speakers
* age between 18 - 65
* normal or corrected to normal vision
* computer and internet access
* fulfill screening criteria of DSM-V for PTSD

Exclusion Criteria:

* Complex PTSD
* Psychotic disorders
* substance dependence or abuse other than nicotine
* Neurological condition
* suicidal ideation or attempt
* change in psychotherapy or pharmacological treatment in the past 3 months.
* Diagnosed/suspected personality Disorder
* Cognitive impairments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Pre to Post improvement of emotion regulatory selection flexibility | Measurements at Baseline and immidiately post treatment
  regulatory selection flexibility is calculated by subtracting adaptive choice from the maladaptive choice specifically by subtracting the proportion of distraction selection in the low intensity stimuli (maladaptive choice) from the proportion of distraction selection in the high intensity stimuli (adaptive choice).
Change from baseline of the total score of the PTSD Checklist (PCL-5) | Measurements at Baseline, immediately post treatment, and 3-months follow-up post treatment
  The PCL-5, is a 20-item PTSD Checklist for DSM-5. Scores can range from 0 to 80, with higher scores reflecting more PTSD symptoms.

OTHER OUTCOMES:
Change from baseline of the total score of the Sheehan Disabilities Scale (SDS) | Measurements at Baseline, immediately post treatment, and 3-months follow-up post treatment
  A composite of three self-rated items measuring the extent to which three domains in participants lives are impaired. Each scale ranges between 0 ("not at all") to 10 ("very much"). The three items are averaged into a single dimensional measure of global functional impairment with scores ranging 0-10.
Change from baseline of the total score of the Beck Depression Inventory (BDI) | Measurements at Baseline, immediately post treatment, and 3-months follow-up post treatment
  A composite score of the 20 items (omitted suicidally item) thus ranging from 0-60
Change from baseline of the total score of the Perceived Ability to Cope With Trauma (PACT) Scale | Measurements at Baseline, immediately post treatment, and 3-months follow-up post treatment
  a 20-item self-report measure of one's beliefs about their capabilities in managing post-trauma sequelae. Two scale scores have been derived: trauma focus (perceived ability to process the trauma), and forward focus (perceived ability to move beyond the trauma). A flexibility score may also be derived, which represents an individual's ability to adaptively use both types of focus.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided